CLINICAL TRIAL: NCT03307876
Title: Intradiscal Injection of an Autologous Alpha-2-macroglobulin (A2M) Concentrate Alleviates Back Pain in FAC-positive Patients
Brief Title: Injection of an Autologous A2M Concentrate Alleviates Back Pain in FAC-positive Patients
Status: Completed | Type: Observational
Sponsor: Scuderi, Gaetano J., M.D. (Other)
Responsible Party: Sponsor
Other Study IDs: 201601
Record Dates: First submitted 2016-06-24; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Low Back Pain
Keywords: biologic,; Alpha 2 Macroglobulin; A2M; back pain; APIC; FAC; FACT
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — lavage sample of the disc for FAC analysis is taken prior to autologous PPP injection. It was discarded after the analysis was complete.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- groups that are fac + and -: autologous PPP injection is given to all patients. Prior to injection, a lavage of the disc space is taken to test for FAC.
  Interventions: Other: autologous PPP injection

INTERVENTIONS:
Other: autologous PPP injection — autologous platelet poor plasma (PPP) injection taken from the participants own blood is injected in to all patients.

SUMMARY:
A cartilage degradation product, the Fibronectin-Aggrecan complex (FAC), has been identified in patients with degenerative disc disease (DDD). Alpha-2-macroglobulin (A2M) can prevent the formation of the G3 domain of aggrecan, reducing the fibronectin-aggrecan G3 complex and therefore may be an efficacious treatment. The present study was designed to determine 1) the ability of autologous concentrated A2M to relieve back pain in patients with LBP from DDD and 2) the ability of FAC to predict the response to this biologic therapy.

24 patients with low back pain and MRI-concordant DDD had prospective evaluation. Oswestry disability index (ODI) and visual analog scores (VAS) were noted at baseline and at 3- and 6-month follow-up. Primary outcome of clinical improvement was defined as patients with both a decrease in VAS of at least 3 points and ODI >20 points. Molecular discography and delayed FAC analysis and injection of platelet poor plasma at the time of the procedure. Patients with FACT-positive assays were significantly more likely to show improvement in their VAS and ODI at follow-up.

DETAILED DESCRIPTION:
Objectives: A cartilage degradation product, the Fibronectin-Aggrecan complex (FAC), has been identified in patients with degenerative disc disease (DDD). Alpha-2-macroglobulin (A2M) can prevent the formation of the G3 domain of aggrecan, reducing the fibronectin-aggrecan G3 complex and therefore may be an efficacious treatment. The present study was designed to determine 1) the ability of autologous platelet poor plasma (PPP) with concentrated A2M to relieve back pain in patients with low back pain (LBP) from DDD and 2) the ability of FAC to predict the response to this biologic therapy.

Study design/setting: Prospective cohort

Patients: 24 patients with low back pain and MRI-concordant DDD

Methods: All patients underwent lavage for molecular discography and delayed FAC analysis and injection of autologous platelet poor plasma (PPP) rich in A2M (Cytonics Autologous Protease Inhibitor Concentrate, APIC) at the time of the procedure. ANOVA with Bonferonni correction for multiple comparisons was performed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater with a history of low back pain complaints primarily dictated by pain with associated sensory symptoms and/or low back pain for 6 months or more who had failed expectant management with NSAIDS, activity modification, and/or physical therapy.
* MRI that demonstrated signs of degenerative disc disease at one or more levels with a Pfirrmann grade of II to IV.
* Age from 18 to 65 with axial back pain of at least 6 months duration.

Exclusion Criteria:

* Patients with a history of oral or injected corticosteroid medication within a three month period prior to disc injection.
* Chronic medical conditions associated with metabolic or inflammatory disorders (insulin-dependent diabetes mellitus, severe coronary artery disease, rheumatic or autoimmune diseases) were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with LBP
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 3 and 6 months
  Change from Baseline ODI at 3 and 6 months

SECONDARY OUTCOMES:
Visual Analogue Score (VAS) | 3 and 6 month
  Change from Baseline VAS at 3 and 6 months

IPD SHARING:
Plan to Share IPD: No